CLINICAL TRIAL: NCT02233504
Title: Pilot Study to Assess Hematologic Response in Patients With Acute Myeloid Leukemia or High Risk Myelodysplastic Syndromes Undergoing Monotherapy With Exjade (Deferasirox)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 40413
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: High Risk MDS or AML Patients
MeSH Terms: interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Exjade® (deferasirox, ICL670)

SUMMARY:
The purpose of this trial is to examine the hematologic response rate of Exjade® in patients with AML and high risk MDS and chronic iron overload from blood transfusions. Deferasirox has been developed as an iron-chelating agent, and unlike deferoxamine, a previously developed iron chelator, deferasirox has the advantage of oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high risk MDS or AML Exjade Pilot Assessing Hematologic Response in AML/MDS UPCC# 40413
* Newly diagnosed acute myeloid leukemia, not a candidate for intensive induction chemotherapy in the judgement of the investigator or unwilling to undergo intensive induction chemotherapy OR
* AML that is refractory or relapsed after treatment with a non-intensive regimen, and not a candidate for allogeneic transplant at this time OR
* MDS, IPSS 1.5 or greater, intolerant or with disease progression/lack of response to hypomethylating agents.
* Age ≥ 18 years and able to provide independent informed consent
* Serum Ferritin: For enrollment on the study: serum ferritin ≥ 500 ng/mL at screening. Samples must be obtained in the absence of concomitant infection. If transfusion is scheduled, draw serum ferritin PRIOR to transfusion.
* ECOG performance status 0-2.
* Sexually active women must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined as amenorrhea for at least 12 months)

Exclusion Criteria:

* Prior therapy with intensive chemotherapy for AML
* Prior therapy with iron chelating agents within the last 6 months.
* Serum creatinine levels greater than 1.5x above the upper limit of normal
* AST or ALT levels greater than 5x the upper limit of normal
* Current therapy for AML or MDS (a ≥ 4 week washout period for any agent used to treat AML or MDS prior to first dose of study drug is required).
* Current therapy with hydrea to control leukocytosis.
* Clinical or laboratory evidence of active Hepatitis B or Hepatitis C (HBsAg in the absence of HBsAb OR HCV Ab positive with HCV RNA positive and ALT above the normal range) infection. In the absence of clinical suspicion for active infection, laboratory testing to assess Hepatitis B or C status will not be required at screening.
* Clinical history of HIV positive test result (ELISA or Western blot). Laboratory testing to assess HIV status will not be required at screening.
* Clinical or self reported history of drug or alcohol abuse within the 12 months prior to enrollment
* ECOG Performance Status > 2
* Uncontrolled systemic hypertension
* Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease not controlled by standard medical therapy
* Clinical diagnosis of or history of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which in the opinion of the investigator would prevent study treatment
* Pregnant or breast feeding women
* Treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days or plan to receive other investigational drugs while participating in the study
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative
* Hematopoietic stem cell transplant for MDS or AML.
* Active CNS leukemia Patients who are found to be ineligible after screening procedures will have the reason for ineligibility documented on the screening log. No further data will be collected in the CRF for these patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10-02 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Mangan, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States